CLINICAL TRIAL: NCT05842655
Title: Digital Technique to Analyze the Wear of Screw-Retained Implant-Supported Metal-Ceramic Dental Prostheses and Natural Tooth as Antagonist. A Pilot Study
Brief Title: Digital Technique to Analyze the Wear of Implants and Natural Tooth as Antagonist.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Principal Investigator, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USAL 2022-AZM
Record Dates: First submitted 2022-12-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Dental Prosthesis Failure
Keywords: Implant supported; morphometry; screw-retained; digital; wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients thats were chosen in order to rehabilitate partial edentulism by dental implants. (Experimental)
  Interventions: Procedure: The wear of screw-retained implant-supported metal-ceramic dental prostheses and natural tooth

INTERVENTIONS:
Procedure: The wear of screw-retained implant-supported metal-ceramic dental prostheses and natural tooth — A novel digital technique to analyze the wear of screw-retained implant-supported metal-ceramic dental prostheses and natural tooth as antagonist

SUMMARY:
The aim of this study was to describe a novel digital technique to analyze the wear of screw-retained implant-supported metal-ceramic dental prostheses and natural tooth as antagonist. Materials and methods: Ten patients were consecutively included to rehabilitate partial edentulism by dental implants. Both the screw-retained implant-supported metal-ceramic dental prostheses and the natural tooth as antagonist were submitted to a digital impression through an intraoral scan to generate a Standard Tessellation Language digital file preoperatively (STL1), at 3 months (STL2), and 6 months (STL3) follow-up. Afterwards, an alignment procedure of the digital files (STL1-STL3) was performed on a reverse engineering morphometric software and volume changes at the screw-retained implant-supported metal-ceramic dental prostheses and the natural tooth as antagonist were analyzed using Student's t-test. Moreover, Gage R&R statistical analysis was conducted to analyze the repeatability and reproducibility of the digital technique.

ELIGIBILITY:
Inclusion Criteria:

* in good health, who presented partial edentulism in the posterior upper maxilla, were consecutively included to rehabilitate partial edentulism by dental implants

Exclusion Criteria:

* all those who do not meet the inclusion criteria

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Wear volume (µm3) of the screw-retained implant-supported metal-ceramic dental prostheses | 3 months follow-up appointment
  Wear volume (µm3) of the screw-retained implant-supported metal-ceramic dental prostheses at 3 months follow-up appointment
Wear volume (µm3) of the screw-retained implant-supported metal-ceramic dental prostheses | 6 months follow-up appointment
  Wear volume (µm3) of the screw-retained implant-supported metal-ceramic dental prostheses at 6 months follow-up appointment
Wear volume (µm3) of the natural tooth as antagonist | 3 months follow-up appointment
  Wear volume (µm3) of the natural tooth as antagonist at 3 months follow-up appointment
Wear volume (µm3) of the natural tooth as antagonist | 6 months follow-up appointment
  Wear volume (µm3) of the natural tooth as antagonist at 6 months follow-up appointment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Castellanos-Cosano L, Rodriguez-Perez A, Spinato S, Wainwright M, Machuca-Portillo G, Serrera-Figallo MA, Torres-Lagares D. Descriptive retrospective study analyzing relevant factors related to dental implant failure. Med Oral Patol Oral Cir Bucal. 2019 Nov 1;24(6):e726-e738. doi: 10.4317/medoral.23082. PMID 31655831
- [Result] Wiley MG. Effects of porcelain on occluding surfaces of restored teeth. J Prosthet Dent. 1989 Feb;61(2):133-7. doi: 10.1016/0022-3913(89)90360-0. PMID 2654359
- [Result] Hudson JD, Goldstein GR, Georgescu M. Enamel wear caused by three different restorative materials. J Prosthet Dent. 1995 Dec;74(6):647-54. doi: 10.1016/s0022-3913(05)80319-1. PMID 8778391
- [Result] Fisher RM, Moore BK, Swartz ML, Dykema RW. The effects of enamel wear on the metal-porcelain interface. J Prosthet Dent. 1983 Nov;50(5):627-31. doi: 10.1016/0022-3913(83)90198-1. PMID 6358468
- [Result] Seghi RR, Rosenstiel SF, Bauer P. Abrasion of human enamel by different dental ceramics in vitro. J Dent Res. 1991 Mar;70(3):221-5. doi: 10.1177/00220345910700031301. PMID 1999562
- [Result] Oh WS, Delong R, Anusavice KJ. Factors affecting enamel and ceramic wear: a literature review. J Prosthet Dent. 2002 Apr;87(4):451-9. doi: 10.1067/mpr.2002.123851. PMID 12011863
- [Result] Ohlmann B, Trame JP, Dreyhaupt J, Gabbert O, Koob A, Rammelsberg P. Wear of posterior metal-free polymer crowns after 2 years. J Oral Rehabil. 2008 Oct;35(10):782-8. doi: 10.1111/j.1365-2842.2008.01865.x. Epub 2008 May 9. PMID 18482349
- [Result] Hmaidouch R, Weigl P. Tooth wear against ceramic crowns in posterior region: a systematic literature review. Int J Oral Sci. 2013 Dec;5(4):183-90. doi: 10.1038/ijos.2013.73. Epub 2013 Oct 18. PMID 24136675
- [Result] Etman MK, Woolford M, Dunne S. Quantitative measurement of tooth and ceramic wear: in vivo study. Int J Prosthodont. 2008 May-Jun;21(3):245-52. PMID 18548965
- [Result] Yilmaz H, Aydin C, Gul BE. Flexural strength and fracture toughness of dental core ceramics. J Prosthet Dent. 2007 Aug;98(2):120-8. doi: 10.1016/S0022-3913(07)60045-6. PMID 17692593
- [Result] Heintze SD, Zellweger G, Sbicego S, Rousson V, Munoz-Viveros C, Stober T. Wear of two denture teeth materials in vivo-2-year results. Dent Mater. 2013 Sep;29(9):e191-204. doi: 10.1016/j.dental.2013.04.012. Epub 2013 Jun 6. PMID 23746749
- [Result] Stober T, Geiger A, Rues S, Dreyhaupt J, Rammelsberg P, Ohlmann B. Factors affecting wear of composite resin denture teeth--24-month results from a clinical study. Clin Oral Investig. 2012 Apr;16(2):413-20. doi: 10.1007/s00784-011-0534-y. Epub 2011 Mar 8. PMID 21384126
- [Result] Zubizarreta-Macho A, Triduo M, Alonso Perez-Barquero J, Guinot Barona C, Albaladejo Martinez A. Novel Digital Technique to Quantify the Area and Volume of Cement Remaining and Enamel Removed after Fixed Multibracket Appliance Therapy Debonding: An In Vitro Study. J Clin Med. 2020 Apr 12;9(4):1098. doi: 10.3390/jcm9041098. PMID 32290554